CLINICAL TRIAL: NCT01891357
Title: A Multicenter Site, Open Label, Phase II Trial to Validate Predictive Markers for the Response Evaluation of a Combined Chemo-immunotherapy in Patients With HER2-positive Early Breast Cancer
Brief Title: Phase II Trial to Validate Markers for a Response Evaluation of a Combined Therapy in Patients With HER2+ Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to significant lack of relevant patient data for evaluation of objectives.
Sponsor: West German Study Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM07 (Neo-PREDICT-HER2); 2012-003679-21 (EudraCT Number)
Record Dates: First submitted 2013-05-14; First posted 2013-07-03 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Ductal, Breast
Keywords: Unilateral primary invasive carcinoma of the breast
MeSH Terms: conditions — Carcinoma, Ductal, Breast | interventions — Pharmaceutical Preparations; Paclitaxel; Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel + Lapatinib + Trastuzumab (Experimental): Paclitaxel 80 mg/m2 weekly for 12 weeks with lapatinib 750 mg P.O. daily and trastuzumab 2 mg/kg IV (loading dose 4 mg/kg) weekly for 12 weeks, biopsy before and after three weeks of study treatment
  Interventions: Procedure: Biopsy before and after three weeks of study treatment; Drug: paclitaxel; Drug: lapatinib; Drug: trastuzumab

INTERVENTIONS:
Procedure: Biopsy before and after three weeks of study treatment — Core biopsies for histological analyses, to be analysed by the central pathology
Drug: paclitaxel
Drug: lapatinib
Drug: trastuzumab

SUMMARY:
The Neo-PREDICT-HER2 Study is phase II trial to validate predictive markers for the response evaluation of a combined chemo-immunotherapy in patients with HER2-positive early breast cancer. The only treatment arm consists of Paclitaxel 80 mg/m2 weekly for 12 weeks with lapatinib 750 mg P.O. daily and trastuzumab 2 mg/kg IV (loading dose 4 mg/kg) weekly for 12 weeks.

DETAILED DESCRIPTION:
Trastuzumab (T)-containing neoadjuvant chemotherapy has been reported to increase the probability of pathological complete response (pCR) in HER2 positive disease up to 67 %. Large trials revealed pCR rates (no remaining invasive and in situ components) of about 30-40 %, if anthracyclines/taxane based polychemotherapy was applied or about 40-45 % if no invasive tumor in the breast and lymph nodes was used as a pCR definition.

Nevertheless, resistance to trastuzumab remains one of the most important challenges in adjuvant and metastatic breast cancer therapy causing poor prognosis with an increased incidence of cerebral metastasis and limited therapeutic options after disease progression6. An improvement shows the combination of trastuzumab and lapatinib, which has been reported to have increased efficacy in in-vitro and in metastatic setting in patients who were mostly resistant to both therapies in the previous course of disease. Recent data from the neoadjuvant setting (neoALTTO) - on a paclitaxel backbone - showed a significantly higher pCR rate after L + T than with either compound separately (47 % vs. 20 % and 27.6 % respectively). Several trials are planned to evaluate the combination of both therapies in the adjuvant and neoadjuvant setting.

Clinical response measured by sequential evaluation of different proliferation markers (such as Ki-67) following a course of neoadjuvant chemotherapy has been demonstrated to correlate significantly with an increased risk of relapse in patients not achieving pathological complete response. It is therefore clinically relevant to evaluate such proliferation tools for early prediction of combination therapy efficacy (chemotherapy and HER2 targeted therapy). So far, it remains unclear which method of proliferation measurement is the optimal marker for response evaluation regarding a combined chemo-immunotherapy. However, measurement of proliferation and apoptosis genes as well as assessment of changes in Phosphatidylinositol 3-kinases (PI3K), Protein Kinase B (AKT), Insulin-like Growth Factor (IGF) and stem cell signalling after a short course of therapy could provide a unique signature for a dynamic response evaluation.

The planned trial will validate predictive markers and a dynamic model based on the sequential evaluation of different proliferation and apoptosis markers. Furthermore it will assess the pCR-rate after 12 weeks of therapy. The aim of the study is to define a predictive marker for the response evaluation of a combined chemo-immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, age at diagnosis 18 - 75 years
2. Histological confirmed unilateral primary invasive carcinoma of the breast
3. Clinical Stage Tumor 1 (cT1) (> 1 cm) - Clinical Stage Tumor 4 (cT4) (if operable, inflammatory breast cancer is excluded)
4. HER2 over-expressing tumor confirmed by: 3+ by Immuno-histochemistry (IHC) and/or HER2/neu gene amplification by fluorescence, chromogenic or silver in-situ hybridization [Fluorescent In-Situ Hybridization (FISH), Chromogenic In-Situ Hybridization (CISH) or Silver In-Situ Hybridization (SISH); > 6 HER2 gene copies per nucleus or a FISH, CISH or SISH test ratio (HER2 gene copies to chromosome 17 signals) of ≥ 2.0]
5. Clinically node positive disease or node negative disease
6. No clinical evidence for distant metastasis (cM0) after conventional staging
7. Performance Status Eastern Cooperative Oncology Group (ECOG) ≤ 1 or Karnofsky Index (KI) ≥ 80%
8. Baseline Left Ventricular Ejection Fraction (LVEF) > 50% measured by echocardiography
9. Negative pregnancy test (urine or serum) within 7 days prior to start of induction treatment in premenopausal patients
10. The patient must be accessible for treatment and follow-up
11. Written informed consent including a written informed consent for shipping of tumor block for central pathology review and evaluation prior to the start of any study procedures

Exclusion Criteria:

1. Known hypersensitivity reaction to the compounds or incorporated substances
2. Known polyneuropathy grade ≥ 2
3. Have acute or currently active or requiring anti-viral therapy hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, stable chronic liver disease per investigator assessment).
4. Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin, pTis of the cervix uteri
5. Prior or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
6. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry
7. Male breast cancer
8. Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
9. Breast feeding women
10. Sequential breast cancer
11. Lack of patient compliance
12. Inadequate organ function including:

    * Leucocytes < 3.5 x 109/l
    * Platelets < 100 x 109/l
    * Absolute Neutrophil Count (ANC) < 1.5 x 109/l
    * Hemoglobin < 9 g/dl
    * Serum Creatinine > 1.5 mg/dl
    * Serum Bilirubin > 1.1 mg/dl
    * Alkaline phosphatase > 2.5 x Upper Limit of Normal (ULN)
    * Aspartate Transaminase (ASAT) and/or Alanine Transaminase (ALAT) > 2.5 ULN
    * Albumin < 2.5 g/dl
13. Uncompensated cardiac function
14. Malabsorption syndrome, disease significantly affecting gastrointestinal function
15. Concomitant use of Cytochrome P450 3A4 (CYP3A4) inhibitors or inducers

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Warm, MD, Principal Investigator — Krankenhaus Köln Holweide
Locations (10):
- Germany (10):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - SLK Kliniken, Heilbronn, Baden-Wurttemberg
  - Klinikum Frankfurt Höchst, Frankfurt am Main, Hesse
  - Niels-Stensen-Kliniken, Georgsmarienhütte, Lower Saxony
  - Krankenhaus Köln Holweide, Brustzentrum, Cologne, North Rhine-Westphalia
  - Klinikum Westfalen GmbH - Knappschaftskrankenhaus, Dortmund, North Rhine-Westphalia
  - Bethesda Krankenhaus, Senologie, Duisburg, North Rhine-Westphalia
  - St. Barbara-KIinik, Hamm, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Praxis für gynäkologische Onkologie am Brustzentrum City, Berlin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients should only have been registered for the study, if final results of screening evaluations were available and all inclusion/exclusion criteria met. This was not true for 3 patients.
  Patients should not have been registered due to distant metastasis. These patients were classified as screening failures and withdrawn from the study.
Groups:
- Paclitaxel + Lapatinib + Trastuzumab: Paclitaxel 80 mg/m2 weekly for 12 weeks with lapatinib 750 mg P.O. daily and trastuzumab 2 mg/kg IV (loading dose 4 mg/kg) weekly for 12 weeks, biopsy before and after three weeks of study treatment
  Biopsy before and after three weeks of study treatment: Core biopsies for histological analyses, to be analysed by the central pathology
  paclitaxel
  lapatinib
  trastuzumab
Period: Overall Study
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Started | 64
Completed | 61
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: ITT: Intent-to-treat population of all randomized patients without screening failures, comprising 61 patients (3 screening failures).
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographics of All Registered Patients
  Participants
    Female | 61
    Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 61

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR)
Description: pCR was defined at the time of surgery and measured by size of residual tumor, proportion of vital cells within invasive carcinoma, number of positive lymph nodes (ypN) and size of the largest lymph node metastasis and ductal carcinoma in situ (ypT). pCR is defined as ypT0/is, ypN0. Further exploratory pCR definitions were ypT0, ypN0 (total pCR) and ypT0/is (near pCR).
Time Frame: Average of 16 weeks
Population: Measurement of pCR: at time of surgery, measured by size of residual tumor, proportion of vital cells per invasive carcinoma, number of positive lymph nodes (ypN), size of largest lymph node metastasis, ductal carcinoma in situ (ypT). Definition of pCR: ypT0/is, ypN0. Exploratory pCR definition: ypT0, ypN0 (total pCR), ypT0/is (near pCR).
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Number analyzed (Participants) | 61
Participants
  ypT0, ypN0 | 19
  ypT0/is | 27
  ypT0/is, ypN0 | 25

2. Secondary Outcome: Event Free Survival (EFS)
Time Frame: 5-year survival
Population: Data were not collected and the outcome cannot be reported
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Time Frame: 5-year survival
Population: Data were not collected and the outcome cannot be reported
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Proliferation and Apoptosis Genes
Description: Proliferation Ki-67, Aurora A Kinase (STK15), survivin, Myb-related protein B (MYBL2),Cyclin B1 and apoptosis genes Bcl2, Epidermal Growth Factor-like 2 (SCUBE2), cleaved caspase C3 will be assessed in the samples from diagnostic and sequential biopsy.
Time Frame: One week before and after three weeks of treatment
Population: Data were not collected and the outcome cannot be reported
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE collection from signature of ICF until end of study per patient, up to 3 years.
Description: Safety population for analysis of toxicities, comprised of 61 patients who were allocated to intervention and received at least one dose of study treatment.
Arm/Group | Paclitaxel + Lapatinib + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 16/61
Other Adverse Events (participants affected / at risk) | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Lapatinib + Trastuzumab (N=61)
Death (Psychiatric disorders) | 1 (1) — suicide
anxiety (Psychiatric disorders) | 1 (1) — Anxiety
Cholecystitis (Gastrointestinal disorders) | 1 (2) — Cholecystitis
Decreased appetite (Gastrointestinal disorders) | 1 (1) — Decreased appetite
Dehydration (Renal and urinary disorders) | 1 (1) — Dehydration
Device related thrombosis (Vascular disorders) | 1 (1) — Device related thrombosis
diarrhoea (Gastrointestinal disorders) | 3 (3) — diarrhoea
Fatigue (General disorders) | 1 (1) — Fatigue
hypokaleamia (Metabolism and nutrition disorders) | 1 (1) — hypokaleamia
impaired healing (Skin and subcutaneous tissue disorders) | 1 (1) — impaired healing
Leukopenia (Blood and lymphatic system disorders) | 1 (1) — Leukopenia
Mucosal Inflammation (Skin and subcutaneous tissue disorders) | 1 (1) — Mucosal Inflammation
Ophthalmic herpes simplex (Eye disorders) | 1 (1) — Ophthalmic herpes simplex
Pneumonia (Infections and infestations) | 1 (1) — Pneumonia
septic shock (Infections and infestations) | 1 (1) — septic shock
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 (1) — Subcutaneous abscess
Syncope (Cardiac disorders) | 1 (1) — Syncope
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Urinary tract infection
Urosepsis (Renal and urinary disorders) | 1 (1) — Urosepsis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel + Lapatinib + Trastuzumab (N=61)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 21 (21) — Blood and lymphatic system disorders
Cardiac disorders (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 (3) — Ear and labyrinth disorders
Eye disorders (Eye disorders) | 5 (5) — Eye disorders
Gastrointestinal disorders (Gastrointestinal disorders) | 59 (133) — Gastrointestinal disorders
General disorders and administration site conditions (General disorders) | 53 (53) — General disorders and administration site conditions
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) — Hepatobiliary disorders
Immune system disorders (Immune system disorders) | 5 (5) — Immune system disorders
Infections and infestations (Infections and infestations) | 30 (30) — Infections and infestations
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 (4) — Injury, poisoning and procedural complications
Investigations (Investigations) | 28 (28) — Investigations
Metabolism and nMetabolism and nutrition disordersutrition disorders (Metabolism and nutrition disorders) | 10 (10) — Metabolism and nutrition disorders
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 12 (12) — Musculoskeletal and connective tissue disorders
Nervous system disorders (Nervous system disorders) | 59 (66) — Nervous system disorders
Psychiatric disorders (Psychiatric disorders) | 15 (15) — Psychiatric disorders
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) — Renal and urinary disorders
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) — Reproductive system and breast disorders
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 31 (31) — Respiratory, thoracic and mediastinal disorders
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 59 (93) — Skin and subcutaneous tissue disorders
Vascular disorders (Vascular disorders) | 14 (14) — Vascular disorders

LIMITATIONS AND CAVEATS:
Only a limited number of core biopsies was available evaluation of dynamic biological changes.

Very slow patient recruitment. Negative study results from ALTTO study did no longer justify further conduct.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days